CLINICAL TRIAL: NCT00452556
Title: The ELDORADO (Eligard®, Docetaxel and Radiotherapy) Study: A Phase II Study of Chemo - Hormonal Therapy and Radiation in High Risk Prostate Cancer
Brief Title: The ELDORADO (Eligard®, Docetaxel and Radiotherapy) Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nova Scotia Cancer Centre (Other)
Responsible Party: Principal Investigator, Derek R Wilke MD,MSc,FRCPC, Research Director, Department of Radiation Oncology, Queen Elizabeth II Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DOCET-L-01892
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Prostatic Neoplasms
Keywords: Prostatic Neoplasms; Radiotherapy; Docetaxel; Leuprolide Acetate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Leuprolide; luprolide acetate gel depot; Radiotherapy, Intensity-Modulated; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Radiotherapy Sequence Arm (Active Comparator): Standard sequence of radiotherapy = whole pelvic lymphatics, proximal seminal vesicles, prostate (or prostate bed) first, then prostate/prostate bed last
  Interventions: Drug: Docetaxel; Drug: Leuprolide Acetate (Eligard®); Radiation: Intensity-Modulated Radiotherapy
- Experimental Radiotherapy Sequence Arm (Experimental): Experimental sequence of radiotherapy = whole pelvic lymphatics, proximal seminal vesicles, prostate (or prostate bed) last, prostate/prostate bed first
  Interventions: Drug: Docetaxel; Drug: Leuprolide Acetate (Eligard®); Radiation: Intensity-Modulated Radiotherapy

INTERVENTIONS:
Drug: Docetaxel — Weekly
  Other Names: Taxotere
Drug: Leuprolide Acetate (Eligard®) — 2.5 years
  Other Names: Androgen deprivation
Radiation: Intensity-Modulated Radiotherapy — Standard sequence = irradiation of pelvic lymphatics, seminal vesicles, and prostate, followed by irradiation of gross tumor (prostate+extraprostatic extension, as determined by MRI)
  Other Names: Radiotherapy
Radiation: Intensity-Modulated Radiotherapy — Experimental sequence = irradiation of pelvic lymphatics, seminal vesicles, and prostate last, irradiation of gross tumor (prostate+extraprostatic extension, as determined by MRI)first
  Other Names: Radiotherapy

SUMMARY:
The purpose of this study is to see if sequence inversion of Intensity - modulated Radiotherapy (IMRT) for prostate cancer, can improve the safety and deliverability of concurrent docetaxel chemotherapy with long - term hormonal therapy. The hypothesis is that inverting the traditional sequence of radiotherapy can delay the time to treatment - induced bowel toxicity.

DETAILED DESCRIPTION:
1.0 Objectives

1.1 Primary objective

To investigate if the inversion of sequencing of multi - phase, intensity - modulated radiotherapy (IMRT), for the treatment of patients with high - risk prostate cancer, can improve the delivery of concurrent, weekly Docetaxel chemotherapy, in concert with long - term androgen deprivation (LTAD).

1.2 Secondary objective

To investigate if the inversion of sequencing of multi - phase IMRT can improve the time to grade 2 or 3 gastrointestinal toxicity, the total amount of Docetaxel that can be delivered, or the quality of life in patients receiving concurrent, weekly Docetaxel chemotherapy, in concert with long - term androgen deprivation (LTAD).

2.0 Background

2.1 Rationale to investigate chemo - radiation in high - risk, non - metastatic prostate cancer

Concurrent chemotherapy and radiotherapy, compared to radiotherapy alone, has resulted in improvements in overall survival and cure in patients with locally advanced head and neck , cervix , and lung cancer . Long - term androgen deprivation (LTAD) and radiotherapy results in modest 10 year overall and biochemical - free relapse rates in patients with "High risk" disease . Treatment intensification, in the form of escalation of radiotherapy dose, the addition of chemotherapy, or the addition of radical prostatectomy, in highly - selected patients, has been proposed in the literature , . Given the success of combining concurrent chemotherapy with radiotherapy in other solid tumor sites, it would seem reasonable to investigate this in patients with high - risk, non - metastatic prostate cancer, as defined in the Canadian consensus document , who are in the worst prognostic category.

2.2 Choice of chemotherapy agent and regimen

The optimal chemotherapy to combine with radiation therapy is unknown for the treatment of prostate cancer. A recent phase III study has, however, shown the superiority of Docetaxel and prednisone chemotherapy over the previous standard regimen, Mitoxantrone and prednisone , in men with metastatic prostate cancer, who demonstrated progression on androgen deprivation. For the first time, an improvement in overall median survival was seen for the regimen containing Docetaxel (18.9 vs 16.5 months, p = 0.009), with 48% of men having a 50% or greater reduction in PSA, and improved HRQOL. Toxicity was felt to be acceptable, with the main toxicities (>30% probability) being: fatigue, alopecia, nausea and/or vomiting, neutropenia, nail changes, sensory neuropathy, and diarrhea. The results of this study were supported by a similar phase III study showing superiority of Docetaxel, estramustine and prednisone over Mitoxantrone and prednisone in patients with progressive, hormone - refractory prostate cancer.

Literature review reveals that there is only one published study of concurrent Docetaxel chemotherapy and external beam radiation. The study by Kumar describes a phase I, dose - escalation study designed to determine the maximum tolerated dose (MTD) of weekly Docetaxel. The patient population included twenty - two patients with localized, "high risk" prostate cancer, and used modern external beam radiotherapy to a conventional dose of 70.2 Gray in 39 fractions, including treatment of the pelvic lymph nodes to a dose of 45 Gray in 25 fractions. They determined that the maximum weekly-tolerated dose of Docetaxel was 20 mg/m2, and that at a dose level of 25 mg/m2, the dose - limiting toxicity was grade 3 diarrhea (using the NCI common toxicity criteria, version 2.0 ), which occurred in 2 patients, necessitating a 25% dose reduction. In addition to clinical feasibility, additional studies suggest that Docetaxel may be a reasonable agent to study. There is evidence from in vitro studies that Docetaxel increases the radio - responsiveness by 2.5 to 3 times , , . Docetaxel inhibits the action of Bcl-2, through the phosphorylation of serine residues on the Bcl-2 molecule, promoting apoptosis via the caspase cascade , a pathway of cell apoptosis also utilized by ionizing radiation. Docetaxel is also felt to inhibit the growth of Bcl-2 negative tumors through overexpression of p27, a protein often lost in androgen - insensitive prostate cancer cells.

A comparison of predictors of radiation and androgen therapy resistance, compared to the dominant targets of docetaxol also highlights why docetaxol may be an ideal agent. A small study by Rossner examined patients who underwent salvage radical prostatectomy after biochemical failure from external beam radiotherapy . Fifty - five percent of patient's salvage radical prostatectomy specimens, that showed viable prostate cancer, demonstrated Bcl-2 overexpression, whereas in a comparison group who underwent radical prostatectomy, matched for known prognostic factors, who had no previous exposure to radiation, there was no detectable Bcl-2 overexpression.

It would also appear that Bcl-2 overexpression is also prognostic for recurrence after radical prostatectomy. In a study by Stackhouse, patients whose radical prostatectomy specimens' demonstrated Bcl-2 overexpression had a 27% versus 69% actuarial probability of relapse - free survival at 100 months, compared to patients whose surgical specimens did not overexpress Bcl-2 (Stackhouse 1999).

In summary, the scientific rationale of using concurrent Docetaxel include: providing biological dose enhancement to tumor cells through radio - sensitization, independent cell kill, aid in the destruction of prostate cancer cells that have radio - resistant phenotypes, and to help overcome cells that have an androgen - insensitive phenotype. It is not anticipated that sufficient drug can be delivered to eradicate distant micro - metastases, therefore we are intentionally targeting patients who are 'high - risk', but not at a very high risk of harboring distant micro - metastases. In personal communication with Dr. Ian Tannock (email correspondence available at request), he supports the idea of weekly, as opposed to every 3 weekly Docetaxel, when the intent is to enhance the efficacy of radiotherapy.

The rationale for utilizing weekly Docetaxel, from a side - effect profile, instead of every 3 weekly Docetaxel, is to avoid the hematological toxicity and Myelosuppression of every 3 weekly Docetaxel, as with weekly administration, myelosuppression is only seen rarely (<3%), even in heavily - pretreated patients with metastatic, hormone - refractory prostate cancer8.

2.3 Rationale for radiotherapy sequence inversion

The standard sequence of radiation therapy portals used to treat prostate cancer, is to treat a large volume first, encompassing regional lymphatics, as well as the primary tumor site, and then treat the prostate, and any local extension of tumor that may be extraprostatic, which is usually a small volume. The major reason is to address all the tumor, both microscopic and grossly evidence tumor, so that areas that harbour tumor do not re - seed an area that has been irradiated, and to prevent progression of tumor. In the case of prostate cancer, the initial radiation portals that encompass the regional lymphatics and prostate also encompass small bowel, large portions of bladder and bone marrow. Whereas IMRT can reduce the volume of small bowel, bladder and bone marrow in the high dose radiation volume, it cannot avoid these organs completely. The smaller volume, which only treats the prostate, can completely avoid the small bowel, largely by treating patients with a full bladder, which pushes the small bowel away from the high dose radiation area. When small bowel, or any organ, can be completely avoided by radiation, it will not result in side effects to that organ.

By treating a small volume first, which avoids small bowel and bone marrow, and knowing that the toxicity of Docetaxel is cumulative, it may be possible to deliver more Docetaxel, in full - doses, without delays, because the small bowel will not be irradiated at the same time as the initiation of Docetaxel, as opposed to the tradition sequence of radiotherapy, where the small bowel will be irradiated at the same time as the initiation of Docetaxel. if the order of the large and boost portals were reversed, as well as, employing IMRT, to sculpt the radiation dose away from the small bowel, for the larger fields.

The reason that a sequence inversion is possible for the treatment of prostate cancer, is that neo - adjuvant and concurrent androgen deprivation results in stasis of prostate cancer cells in the radiation volumes, so that there is virtually no added risk of prostate cancer cells migrating from the pelvic lymphatics while the prostate is being irradiated.

2.4 Overlapping treatment - related toxicities and rationale for sequence inversion

The anticipated dose - limiting acute toxicity, common to both modalities is, treatment - related diarrhea. A recent study by Ashman retrospectively examined 27 patients who underwent whole pelvic radiotherapy using 2D, 3D conformal techniques and IMRT. Overall, 9 patients (33%) experienced acute Grade 2 gastrointestinal toxicity, and only 1 of these patients was treated with IMRT. Antidiarrheal medication was required for 6 patients (22%). However, 5 of these 6 patients also received chemotherapy (either concurrent vinblastine/estramustine or neoadjuvant carboplatin, estramustine and paclitaxel, breakdown by chemotherapy regiment not specified in publication), and none were treated with IMRT. No Grade 3 or higher acute or late GI toxicities were observed. No cases of late radiation enteritis were observed.

ELIGIBILITY:
Inclusion Criteria:

* A histological diagnosis of adenocarcinoma of the prostate
* Life expectancy greater than 5 years.
* ECOG performance status < 1.
* Signed, written informed consent prior to randomization.
* Any one, or more, of the following criteria:

  * TNM stage T2c, T3a or T3b
  * Gleason score 8 to 10, as determined by central institutional review.
  * PSA > 20 mcg/L, but < 50 mcg/L. OR Have a > 50% chance of recurrence after radical prostatectomy, as predicted by the Kattan Nomogram and
  * Post - op PSA < 1.0 mcg/L.
  * Must be able to start protocol treatment within 6 months from date of surgery.
* No evidence of metastasis, as determined by bone scan and Chest x-ray/CT abdomen/pelvis.
* Adequate marrow reserve and end - organ function

  * Leukocytes > 3,000/mcL.
  * Absolute neutrophil count > 1,500/mcL
  * Platelets > 100,000/mcL
  * Total bilirubin < 1.2 x upper limit of normal for the institution.
  * AST(SGOT)/ALT(SGPT) greater than 1.5 X institutional upper limit of normal
  * Creatinine within normal institutional limits OR
  * Creatinine clearance > 60 mL/min using the Crockfort - Gault formula for patients with creatinine levels above institutional normal.

Exclusion Criteria:

* PSA > 50 µg/L.
* Previous pelvic radiotherapy
* Sensitivity to Docetaxel chemotherapy.
* Grade 2 or greater NCI CTCAE version 3.0 neuropathy.
* Prior malignancy within the last 5 years, other than prostate cancer, except:

  * Patients with adequately treated non - melanoma cutaneous malignancies.
  * Patients with a history of a curatively treated malignancy (including patients with superficial bladder cancer) who have not had evidence of recurrence for a minimum of 5 years.
* Patients with a history of hypersensitivity to polysorbate 80.
* Patients with a known history of viral hepatitis (B,C).

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2007-05; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
To investigate if the inversion of sequencing of multi - phase, intensity - modulated radiotherapy (IMRT), for the treatment of patients with high - risk prostate cancer, can improve the delivery of concurrent, weekly Docetaxel chemotherapy, in conc | 3 years

SECONDARY OUTCOMES:
To investigate if the inversion of sequencing of multi - phase IMRT can improve the time to grade 2 or 3 gastrointestinal toxicity. | 3 years
total amount of Docetaxel that can be delivered | 3 years
quality of life in patients receiving concurrent, weekly Docetaxel chemotherapy, in concert with long - term androgen deprivation (LTAD). | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Derek R Wilke, MD,MSc,FRCPC, Principal Investigator — Nova Scotia Cancer Centre, Department of Radiation Oncology, Dalhousie University
Locations (1):
- Nova Scotia Cancer Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Wilke D, Wood L, Cwajna S, Rutledge R, Hollenhorst H, Bowes D, Patil N, Ago CT, Pignol JP. Sequence Inversion to Facilitate Concurrent Radiotherapy and Systemic Therapy. A Proof of Principle Study in the Setting of a Phase II Randomized Trial in Prostate Cancer. Front Oncol. 2020 Sep 30;10:570660. doi: 10.3389/fonc.2020.570660. eCollection 2020. PMID 33102224